| 1 | Official Title: "Does Intravenous Lactated Ringer's Solution Raise |
|----|--------------------------------------------------------------------|
| 2 | Serum Lactate?" |
| 3 | |
| 4 | NCT number: NCT02950753 |
| 5 | |
| 6 | Date approved by IRB: Nov 17, 2016 |
| 7 | |
| 8 | |
| 9 | |
| 10 | |
| 11 | |
| 12 | |
| 13 | |
| 14 | |
| 15 | |
| 16 | |
| 17 | |
| 18 | |
| 19 | |
| 20 | |
| 21 | |
| 22 | |
| 23 | |

## **Introduction**

24

45

46

25 26 Since "early goal-directed therapy," early recognition of septic shock using the serum 27 lactate has become standard of care [1-4]. Indeed, the central place of lactate in sepsis 28 care has been promoted by the Surviving Sepsis campaign, and it is now backed by 29 financial incentives for hospitals with its adoption as a CMS Core Measure [5]. 30 31 In this context, it is important to elucidate all possible causes of hyperlactatemia. 32 Previous studies have shown that serum lactate increases in all shock states, not just 33 septic shock [6]. Furthermore, lactate has also been shown to increase from albuterol [7], 34 anti-retroviral medications, metformin, propofol, and alcohols [8]. 35 36 According to Surviving Sepsis Guidelines, patients diagnosed with septic shock should 37 receive 30 mL/kg of crystalloid solution within three hours [9]. One commonly used 38 crystalloid, Lactated Ringer's solution (LR), contains 28 mmol/L of racemic lactate in the 39 form of sodium lactate. While lactate is rapidly metabolized by the liver and kidney, 40 aggressive fluid resuscitation with LR may transiently raise serum lactate, potentially 41 confounding the interpretation of this test. 42 43 There has only been one trial looking at the question of whether administration of LR 44 raises serum lactate. That study did not show a difference in lactate levels in those

receiving LR versus those receiving alternative crystalloid solutions. However, that study

used only 1 liter of LR delivered over one hour [10]. As mentioned above, patients in

septic shock are mandated to receive 30 mL/kg of crystalloid solution, and the fluids are typically given at a rate faster than 1 liter per hour. Therefore, when LR is given at a volume and rate more similar to what is done for septic shock patients, LR may have an effect on serum lactate level that was not identified in the previous study. Thus, we propose a double-blind, randomized controlled trial to investigate whether the administration of intravenous LR at 30 mL/kg increases levels of serum lactate. As our study compares the effect of NS and LR, it lends itself easily to secondarily investigating changes in sodium (Na), chloride (Cl), and pH in the NS group compared to the LR group. **Materials and Methods Study Design and Setting** 

volunteers, made up primarily of family, friends, and colleagues of the investigators.

All subjects will be healthy volunteers aged 18 years or older. Healthy volunteers are

defined as subjects with no acute symptoms who meet none of the following exclusion

This will be a double-blind, randomized controlled trial performed on a group of healthy

overload (congestive heart, renal, or hepatic failure), baseline serum lactate level >2.2

criteria: pregnant, breast-feeding, prisoners, history of conditions associated with fluid

mmol, and baseline creatinine >1.5 mg/dL.

47

48

49

50

51

52

53

54

55

56

57

58

59

60

61

62

67

68

69

70 71 All volunteers will fill out a short data collection form assessing their age, weight, 72 gender, and medical history. All volunteers will signed a written consent, approved by the 73 IRB. 74 75 A random-number generator will be used to assign each subject to either LR or NS. After 76 assignment, a pharmacist with no role in data collection prepared the fluids in a locked 77 room. The pharmacist will use an opaque black bag to obscure the fluids. The subjects 78 will then receive 30 mL/kg rounded to the nearest 100 mL of the solution to which they 79 were randomized. 80 81 An investigator will place an 18 gauge IV in one upper extremity, and an initial serum 82 lactate and electrolyte panel will be drawn, measured using the i-STAT 1 analyzer 83 (Abbott Point of Care, Princeton, NJ). Fluids will be administered as a rapid bolus via 84 pressure bag. Post-treatment blood will be drawn from the contralateral upper extremity 85 five minutes after the conclusion of the IV fluid administration. 86 87 **Outcomes** 88 89 The primary outcome will be the difference in change in serum lactate levels between the 90 LR and NS groups. Secondarily, we will compare the change in lactate within each group 91 (before and after treatment), and we will compare the change in pH, creatinine, 92 bicarbonate, Na, and Cl levels between NS and LR groups.

| O | 2 |
|---|---|
| フ | ) |

94

## **Data Analysis**

95

We powered the study as follows. A sample size of 30 achieves 80% power to detect a
difference of 0.5 mmol/L in the mean change in lactate between the NS and LR groups
assuming a standard deviation of differences of 0.5 and an alpha of 0.05. We chose the
value of 0.5 mmol/L by clinical gestalt based on what we consider a clinically significant
difference in lactate levels. Before and after treatment lactate levels will be compared
within each group using paired t-tests. We will compare the change in mean lactate and
the change in other variables (pH, creatinine, bicarbonate, Na, and Cl) between the LR

104

105

103

## References

- 1. Rivers E, Nguyen B, Havstad S, et al. Early goal-directed therapy in the treatment of
- severe sepsis and septic shock. *N Engl J Med*. 2001; 345 (19): 1368–77.
- 108 2. Process Investigators, Yealy DM, Kellum JA, et al, A randomized trial of protocol-
- based care for early septic shock. N Engl J Med. 2014;370:1683–1693.
- 3. Mouncey PR, Osborn TM, Power GS, et al. Trial of early, goal-directed resuscitation
- 111 for septic shock. *N Engl J Med*. 2015;372:1301–1311.

and NS groups using two-tailed t-tests.

- 4. ARISE Investigators, Anzics Clinical Trials Group, Peake SL, et al. Goal-directed
- resuscitation for patients with early septic shock. *N Engl J Med.* 2014;371:1496–1506.
- 5. Centers for Medicare & Medicaid Services. CMS specifications manual version 5.2a.
- 115 Available at:

- 116 <a href="https://www.qualitynet.org/dcs/ContentServer?c=Page&pagename=QnetPublic%2FPage">https://www.qualitynet.org/dcs/ContentServer?c=Page&pagename=QnetPublic%2FPage</a>
- 117 <u>%2FQnetTier3&cid=1228775749207</u>. Accessed August 22, 2017
- 6. Cecconi M., De Backer D., Antonelli M, et al. Consensus on circulatory shock and
- hemodynamic monitoring. Task force of the European Society of Intensive Care
- 120 Medicine. *Intensive Care Med.* 2014; 40:1795–815.
- 7. Zitek T, Cleveland N, Rahbar A, et al. Effect of Nebulized Albuterol on Serum Lactate
- and Potassium in Healthy Subjects. Acad Emerg Med. 2016; 23(6):718-21.
- 8. Kraut, JA. Madias NE. Lactic Acidosis. *N Engl J Med.* 2014;371:2309-19.
- 9. Dellinger R, Levy M, Rhodes A, et al. Surviving Sepsis Campaign: international
- guidelines for the management of severe sepsis and septic shock 2012. Crit Care Med.
- 126 2013; 41: 580–637.
- 127 10. Didwania A, Miller J, Kassel D, et al. Effect of intravenous lactated Ringer's solution
- infusion on the circulating lactate concentration: Part 3. Results of a prospective,
- randomized, double-blind, placebo-controlled trial. Crit Care Med. 1997; 25(11):1851-4.

130